CLINICAL TRIAL: NCT03712007
Title: Comparison of Two Miniscrew Anchored Maxillary Protraction Protocols: a Randomized Clinical Trial
Brief Title: Comparison of Two Miniscrew Anchored Maxillary Protraction Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Felicia Miranda, DDS, MSc. and PhD Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 67610717.7.0000.5417
Record Dates: First submitted 2018-10-07; First posted 2018-10-19 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Malocclusion, Angle Class III; Crossbite (Anterior) (Posterior)
Keywords: Orthodontic Anchorage Procedures; Malocclusion, Angle Class III; Palatal Expansion Technique.; Cone-Beam Computed Tomography; Dental Models
MeSH Terms: conditions — Malocclusion, Angle Class III; Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAMP therapy with MARPE expander (Experimental): The experimental group will comprise 20 patients submitted to miniscrew anchored maxillary protraction (MAMP) with a tooth-bone-borne expander as anchorage in the maxillary arch. The miniscrew assisted rapid palatal expander (MARPE) will be used.
  Interventions: Device: MAMP therapy with MARPE expander
- MAMP therapy with Hyrax expander (Active Comparator): The active comparator group will comprise 15 patients submitted to miniscrew anchored maxillary protraction (MAMP) with a tooth-borne expander as anchorage in the maxillary arch. The conventional hyrax expander will be used.
  Interventions: Device: MAMP therapy with Hyrax expander

INTERVENTIONS:
Device: MAMP therapy with MARPE expander — Twenty patients will be submitted to MAMP therapy with MARPE expander as anchorage in the maxillary arch. The appliance anchorage will be provided by bands adapted on the maxillary first permanent molars and circumferential clamps in the maxillary canines or premolars. The maxillary and mandibular miniscrews will be placed in the same section. After a 24-hour period, parents will be oriented to activate the expander screw. Patients will be instructed to wear intermaxillary elastics connecting the maxillary first molar hooks to the mandibular mini-implants.
  Arms: MAMP therapy with MARPE expander
Device: MAMP therapy with Hyrax expander — Fifteen patients will be submitted to MAMP therapy with Hyrax expander as anchorage in the maxillary arch. The appliance anchorage will be provided by bands adapted on the maxillary first permanent molars and circumferential clamps in the maxillary canines or premolars. The mandibular miniscrews will be placed and after a 24-hour period, parents will be oriented to activate the expander screw. Patients will be instructed to wear intermaxillary elastics connecting the maxillary first molar hooks and the mandibular mini-implants.
  Arms: MAMP therapy with Hyrax expander

SUMMARY:
This study evaluates the dentoskeletal effects produced by two maxillary protraction protocols in adolescent patients. Half of participants will be treated with a tooth-borne and tooth-bone-borne expanders as anchorage in the maxillary arch. Miniscrews will be used as anchorage in the mandibular arch for both groups.

DETAILED DESCRIPTION:
Class III malocclusion treatment in growing patients is challenging. A new treatment for maxillary protraction using skeletal anchorage reported an efficient maxillary protraction in the late mixed dentition an early permanent dentition. Therefore, the aim of this study is to compare the dentoskeletal effects produced by two maxillary protraction protocols anchored on miniscrews.

The sample will be recruited at the Orthodontic Clinic of Bauru Dental School, University of São Paulo, Brazil. A sample of thirty-five patients, between 9 and 13 years old will be selected. The inclusion criteria are: Class III malocclusion associated with anterior crossbite. The participants will be allocated into 2 groups. Group 1 will comprise 20 individuals treated with a tooth-bone-borne expander and 2 miniscrews in the mandible Group 2 will comprise 15 individuals treated with a tooth-borne expander and 2 miniscrews in the mandible. Digital models and cone-beam computed tomography (CBCT) will be obtained before (T1) and 12 months after treatment (T2). Occlusal radiographs and partial (canine to canine) models will be obtained before and immediately after expansion. Two-dimensional cephalometric evaluations will be performed in the Dolphin® software. The arch width, arch perimeter and arch length will be analyzed with the Orthoanalyzer® software. Three-dimensional superimposition at the cranial base of T1 and T2 CBCT images will be performed. The inter incisor diastema will be evaluated by occlusal radiographs and dental models. Discomfort, pain and quality of life will evaluated by questionnaires. After verifying the normal distribution, the intragroup comparison will be performed with paired t test and intergroup comparison will be performed with t test. In the case of lost to follow-up patients, intention to treat analysis will be used. A significance level of 5% will be regarded for all tests.

Temporary pain and discomfort are possible after the installation of the miniscrews. Patients and legal guardians will be informed. After the consent, the treatment can be stoped at any time.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes;
* Ages ranging from 9 to 13 years old;
* Class III malocclusion;
* Mandibular canines erupted.

Exclusion Criteria:

* Previous orthodontic treatment;
* Cleft lip and palate;
* Craniofacial syndromes;
* Systemic and/or neurological diseases.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Maxillary sagittal skeletal discrepancy | 12 months
  CBCT exams will be obtained before (T1) and after treatment (T2). Reformatted lateral cephalometric images will be obtained using Dolphin software for comparisons with conventional cephalograms. The maxillary sagittal skeletal discrepancy will be observed using the variables: SNA, Co-A, Condylion to ANS and others.
Mandibular sagittal skeletal discrepancy | 12 months
  CBCT exams will be obtained before (T1) and after treatment (T2). Reformatted lateral cephalometric images will be obtained using Dolphin software for comparisons with conventional cephalograms. Mandibular sagittal skeletal discrepancy will be observed using the variables: Co-Gn, SNB, Gonial/Jaw Angle and others.
Vertical skeletal discrepancy | 12 months
  CBCT exams will be obtained before (T1) and after treatment (T2). Reformatted lateral cephalometric images will be obtained using Dolphin software for comparisons with conventional cephalograms. Vertical skeletal discrepancy will be observed using the variables: Occ Plane to SN, NF - FH (PP-FH), SN - GoGn, SN- Palatal Plane and others.
Teeth discrepancy | 12 months
  CBCT exams will be obtained before (T1) and after treatment (T2). Reformatted lateral cephalometric images will be obtained using Dolphin software for comparisons with conventional cephalograms. Teeth discrepancy will be observed using the variables: Overjet, Overbite, Interincisal Angle (U1-L1), Molar Relation, Mesial Molar Relationship, U1 - Palatal Plane, IMPA and others.
Soft tissue discrepancy | 12 months
  CBCT exams will be obtained before (T1) and after treatment (T2). Reformatted lateral cephalometric images will be obtained using Dolphin software for comparisons with conventional cephalograms. Soft tissue discrepancy will be observed using the variables: Nasolabial Angle (Col-Sn-UL), Upper Lip to E-Plane, Lower Lip to E-Plane, Upper Lip - S line, Lower Lip - S line and others.

SECONDARY OUTCOMES:
Maxillary and mandibular inter-first permanent molar distances | 12 months
  Arch dimensions will be measured in digital dental models obtained before (T1) and after treatment (T2).
Maxillary and mandibular intercanine distances | 12 months
  The intercanine distance will be measured in digital dental models obtained before (T1) and after treatment (T2).
Maxillary and mandibular dental arches perimeters | 12 months
  Arch perimeter will be measured in digital dental models obtained before (T1) and after treatment (T2).
Maxillary and mandibular dental arches lengths | 12 months
  Arch lenght will be measured in digital dental models obtained before (T1) and after treatment (T2).
Inclination of maxillary and mandibular first permanent molars | 12 months
  Teeth inclination will be measured in digital dental models obtained before (T1) and after treatment (T2).
Amount of interincisor diastema | 7 days
  The interincisor diastema will be measured in the occlusal radiograph and partial model obtained immediately after expansion.
Three-dimensional changes | 12 months
  Three-dimensional changes will be observed by the cranial base superimposition of the CBCT exams obtained before (T1) and after treatment (T2).
Discomfort and pain | 1 month
  Discomfort and pain will be evaluated using a visual analog scale of 10-cm, where 0-cm is no discomfort/pain and 10-cm is the greatest discomfort/pain.
Parents perception of pain | 1 month
  Parents perception of pain will be evaluated using a visual analog scale of 10-cm, where 0-cm is no discomfort/pain and 10-cm is the greatest discomfort/pain.
Quality of life evaluation | 12 months
  CPQ (Child Perceptions Questionnaires) will be used to evaluated quality of life. The CPQ8-10 and CPQ11-14 will be applied before (T1), during and after (T2) treatment for patients of both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miranda F, Cunha Bastos JCD, Magno Dos Santos A, Janson G, Pereira Lauris JR, Garib D. Dentoskeletal comparison of miniscrew-anchored maxillary protraction with hybrid and conventional hyrax expanders: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2021 Dec;160(6):774-783. doi: 10.1016/j.ajodo.2021.02.017. Epub 2021 Sep 9. PMID 34509329
- [Derived] Miranda F, Garib D, Pugliese F, da Cunha Bastos JC, Janson G, Palomo JM. Upper airway changes in Class III patients using miniscrew-anchored maxillary protraction with hybrid and hyrax expanders: a randomized controlled trial. Clin Oral Investig. 2022 Jan;26(1):183-195. doi: 10.1007/s00784-021-03989-3. Epub 2021 May 27. PMID 34041608